CLINICAL TRIAL: NCT01852188
Title: A Comparison of Sterile and Non-sterile Gloves for the Incidence of Chorioamnionitis During Labor: a Randomized Controlled Trial
Brief Title: Intrapartum Study of Sterile and Clean Gloves
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HR 20638
Record Dates: First submitted 2012-04-18; First posted 2013-05-13 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Chorioamnionitis
Keywords: Intrapartum; Glove; Chorioamnionitis
MeSH Terms: conditions — Chorioamnionitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nonsterile (Other): Patients will be randomized to either sterile or clean gloves during intrapartum vaginal exams.
  Interventions: Other: Type of glove used for intrapartum vaginal exams
- Sterile (Other): Patients will be randomized to either sterile or clean gloves during intrapartum vaginal exams.
  Interventions: Other: Type of glove used for intrapartum vaginal exams

INTERVENTIONS:
Other: Type of glove used for intrapartum vaginal exams — Patients will be randomized to either sterile or clean gloves during intrapartum vaginal exams.

SUMMARY:
The purpose of this study is to determine whether the use of sterile or clean gloves during labor exams affects the rate of chorioamnionitis. Chorioamnionitis is an infection of the membranes around the baby.

DETAILED DESCRIPTION:
The importance of this study is that intrapartum vaginal exams (while patients are laboring) are performed routinely in modern obstetrical practice, and there is no randomized trial available assessing the relationship between the type of glove used and the rate of chorioamnionitis.

ELIGIBILITY:
Inclusion Criteria:

* Spontaneous or induced labor
* Rupture of membranes < 12 hours
* Nulliparous or multiparous
* Gestational age greater than or equal to 34 weeks
* Age greater than or equal to 18

Exclusion Criteria:

* Contraindications to labor
* Multiple gestations
* Rupture of Membranes greater than 12 hours
* Gestational age less than 34 weeks
* Non-English speaking patients

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2011-05 (Actual); Primary Completion 2014-11-02 (Actual); Study Completion 2014-11-02 (Actual)

PRIMARY OUTCOMES:
Clinical chorioamnionitis | participants will be followed during their intrapartum hospital stay, an expected average of 48-72hrs
  Clinical chorioamnionitis with at least two of the four criteria met-maternal fever of 38 degrees Celsius or greater, maternal tachycardia (pulse >100), fetal tachycardia (fetal heart rate >160), and/or fundal tenderness

CONTACTS AND LOCATIONS:
Overall Officials: Laura Houston, MD, Principal Investigator — Medical University of South Carolina; Donna Johnson, Study Chair — Medical University of South Carolina, Obstetrics-Gynecology
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States